CLINICAL TRIAL: NCT02674854
Title: A Prospective, Double-masked, Randomized, Multi-center, Active Controlled, Parallel-group, 3-month Study Assessing the Safety and Ocular Hypotensive Efficacy of PG324 Ophthalmic Solution Compared to AR-13324 Ophthalmic Solution 0.02% and Latanoprost Ophthalmic Solution 0.005% in Subjects With Elevated Intraocular Pressure
Brief Title: Double-masked Study of PG324 Ophthalmic Solution in Patients With Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG324-CS302
Record Dates: First submitted 2016-02-01; First posted 2016-02-05 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — netarsudil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PG324 Ophthalmic Solution 0.02%/0.005% (Experimental): Fixed combination of netarsudil 0.02%, latanoprost 0.005 % ophthalmic solution
  Interventions: Drug: PG324 Ophthalmic Solution 0.02%/0.005%
- Netarsudil (AR-13324) ophthalmic solution 0.02% (Active Comparator): Netarsudil 0.02% ophthalmic solution
  Interventions: Drug: Netarsudil (AR-13324) ophthalmic solution 0.02%
- Latanoprost ophthalmic solution 0.005% (Active Comparator): Latanoprost 0.005 % ophthalmic solution
  Interventions: Drug: Latanoprost ophthalmic solution 0.005%

INTERVENTIONS:
Drug: PG324 Ophthalmic Solution 0.02%/0.005% — 1 drop daily in the evening (PM) in both eyes (OU)
  Arms: PG324 Ophthalmic Solution 0.02%/0.005%
Drug: Netarsudil (AR-13324) ophthalmic solution 0.02% — 1 drop daily in the evening (PM) in both eyes (OU)
  Arms: Netarsudil (AR-13324) ophthalmic solution 0.02%
Drug: Latanoprost ophthalmic solution 0.005% — 1 drop daily in the evening (PM) in both eyes (OU)
  Arms: Latanoprost ophthalmic solution 0.005%

SUMMARY:
To evaluate ocular hypotensive efficacy and safety of PG324 Ophthalmic Solution compared to netarsudil (AR-13324) ophthalmic solution 0.02% and latanoprost ophthalmic solution 0.005%

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older (19 years of age or older in Canada)
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension(OHT) in both eyes
3. Unmedicated intraocular pressure >20mmHg and <36mmHg in both eyes at 2 qualification visits
4. Best corrected visual acuity (BCVA) equivalent to 20/200 Snellen or better
5. Able to give informed consent and follow study instructions

Exclusion Criteria:

Ophthalmic:

1. Clinically significant ocular disease
2. Pseudoexfoliation or pigment dispersion component glaucoma, history of angle closure or narrow angles
3. Unmedicated intraocular pressure ≥36mmHg in either eye or use of more than 2 ocular hypotensive medications within 30 days of screening
4. Known hypersensitivity to any component of the formulation or latanoprost
5. Previous glaucoma surgery or refractive surgery
6. Ocular trauma within 6 months prior to screening
7. Any ocular surgery or non-refractive laser treatment within 3 months prior to screening
8. Recent or current ocular infection or inflammation in either eye
9. Use of ocular medication in either eye of any kind within 30 days of screening and throughout of the study
10. Mean central corneal thickness >620µm at screening in either eye
11. Any abnormality preventing reliable applanation tonometry of either eye

    Systemic:
12. Clinically significant abnormalities in lab tests at screening
13. Clinically significant systemic disease
14. Participation in any investigational study within 60 days prior to screening
15. Systemic medication that could have had a substantial effect on IOP within 30 days prior to screening, or anticipated to be used during the study
16. Women of childbearing potential who were pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2016-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, MBA, Study Director — Aerie Pharmaceuticals, Inc.
Locations (1):
- Aerie Pharmaceuticals, Bedminster, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Walter TR, Ahmed IK et al. Ophthalmology glaucoma, 2019, pg. 1-10 https://doi.org/10.1016/j.ogla.2019.03.007
- [Derived] Asrani S, Bacharach J, Holland E, McKee H, Sheng H, Lewis RA, Kopczynski CC, Heah T. Fixed-Dose Combination of Netarsudil and Latanoprost in Ocular Hypertension and Open-Angle Glaucoma: Pooled Efficacy/Safety Analysis of Phase 3 MERCURY-1 and -2. Adv Ther. 2020 Apr;37(4):1620-1631. doi: 10.1007/s12325-020-01277-2. Epub 2020 Mar 12. PMID 32166538
- [Derived] Wisely CE, Sheng H, Heah T, Kim T. Effects of Netarsudil and Latanoprost Alone and in Fixed Combination on Corneal Endothelium and Corneal Thickness: Post-Hoc Analysis of MERCURY-2. Adv Ther. 2020 Mar;37(3):1114-1123. doi: 10.1007/s12325-020-01227-y. Epub 2020 Jan 24. PMID 31981106

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PG324 Ophthalmic Solution 0.02%/0.005% | Netarsudil (AR-13324) Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
Started | 245 | 255 | 250
Completed | 221 | 228 | 236
Not Completed | 24 | 27 | 14
Not completed — Adverse Event | 17 | 15 | 5
Not completed — Withdrawal by Subject | 1 | 5 | 4
Not completed — No-compliant subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Lack of Efficacy | 0 | 3 | 0
Not completed — Disallowed Concurrent Medication | 2 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Subject missed V6.2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PG324 Ophthalmic Solution; Netarsudil (AR-13324) Ophthalmic Solution 0.02%; Latanoprost Ophthalmic Solution 0.005%: 1 drop daily in the evening (PM) in both eyes (OU)
- Total: Total of all reporting groups
Arm/Group | PG324 Ophthalmic Solution | Netarsudil (AR-13324) Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005% | Total
Number analyzed (Participants) | 245 | 255 | 250 | 750
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 118 | 109 | 112 | 339
  >=65 years | 127 | 146 | 138 | 411
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.81) | 64.5 (10.58) | 64.3 (11.41) | 64.3 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 153 | 144 | 449
  Male | 93 | 102 | 106 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 48 | 55 | 148
  Not Hispanic or Latino | 200 | 207 | 195 | 602
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 7 | 11 | 6 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 74 | 76 | 79 | 229
  White | 161 | 165 | 163 | 489
  More than one race | 2 | 3 | 0 | 5
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Mean intraocular pressure(IOP) at 08:00, 10:00 and 16:00 hours, at Day 15, Day 43 and Day 90, as measured by Goldmann applanation tonometry.
Time Frame: 3 months
Population: Intent to treat (ITT) population with Monte Carlo Markov Chain (MCMC) imputation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PG324 Ophthalmic Solution | Netarsudil (AR-13324) Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 245 | 255 | 250
mmHg
  Day 1, 0800 hours | 24.69 (3.422) | 24.66 (3.148) | 24.75 (3.240)
  Day 1, 1000 hours | 23.33 (3.399) | 23.40 (3.538) | 23.23 (3.339)
  Day 1, 1600 hours | 22.37 (3.492) | 22.76 (3.558) | 22.59 (3.451)
  Day 15, 0800 hours | 16.06 (3.370) | 19.35 (4.279) | 18.10 (3.375)
  Day 15, 1000 hours | 15.31 (3.272) | 17.99 (3.909) | 17.61 (3.264)
  Day 15, 1600 hours | 15.16 (3.032) | 17.53 (3.772) | 17.08 (3.283)
  Day 43, 0800 hours | 16.43 (3.717) | 19.52 (4.273) | 17.93 (3.586)
  Day 43, 1000 hours | 15.54 (3.533) | 18.40 (3.810) | 17.35 (3.224)
  Day 43, 1600 hours | 15.45 (3.525) | 17.95 (3.776) | 17.09 (3.271)
  Day 90, 0800 hours | 16.45 (3.572) | 19.72 (4.419) | 17.98 (3.400)
  Day 90, 1000 hours | 15.58 (3.307) | 18.30 (3.846) | 17.48 (3.366)
  Day 90, 1600 hours | 15.52 (3.210) | 17.94 (3.627) | 17.14 (3.044)
Statistical Analysis 1: Comparison: PG324 Ophthalmic Solution vs Netarsudil (AR-13324) Ophthalmic Solution 0.02%; Test type: Superiority; p < 0.0001, t-test, 2 sided; PG324 vs. netarsudil
Statistical Analysis 2: Comparison: PG324 Ophthalmic Solution vs Latanoprost Ophthalmic Solution 0.005%; Test type: Superiority; p < 0.0001, t-test, 2 sided; PG324 vs. latanoprost

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the 90 day treatment period.
Description: Safety population, defined as all randomized subjects who received at least 1 dose of investigational product. One subject was randomized to PG324 ophthalmic solution; however, the subject received latanoprost ophthalmic solution 0.005%, resulting in 1 less subject counted in the safety population for PG324 ophthalmic solution and 1 additional subject in the safety population for latanoprost ophthalmic solution 0.005% relative to the numbers in the respective randomized populations
Arm/Group | PG324 Ophthalmic Solution | Netarsudil (AR-13324) Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
All-Cause Mortality (participants affected / at risk) | 0/244 | 1/255 | 0/251
Serious Adverse Events (participants affected / at risk) | 2/244 | 6/255 | 5/251
Other Adverse Events (participants affected / at risk) | 157/244 | 143/255 | 78/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG324 Ophthalmic Solution (N=244) | Netarsudil (AR-13324) Ophthalmic Solution 0.02% (N=255) | Latanoprost Ophthalmic Solution 0.005% (N=251)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Vertebral Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG324 Ophthalmic Solution (N=244) | Netarsudil (AR-13324) Ophthalmic Solution 0.02% (N=255) | Latanoprost Ophthalmic Solution 0.005% (N=251)
Conjunctival Hyperaemia (Eye disorders) | 126 (126) | 102 (102) | 51 (51)
Cornea Verticillata (Eye disorders) | 32 (32) | 25 (25) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 14 (14) | 17 (17) | 2 (2)
Corneal Disorder (Eye disorders) | 14 (14) | 12 (12) | 0 (0)
Instillation Site Pain (General disorders) | 42 (42) | 23 (23) | 15 (15)
Instillation Site Discomfort (General disorders) | 15 (15) | 16 (16) | 2 (2)
Vital Dye Staining Cornea Present (Investigations) | 8 (8) | 13 (13) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT02674854/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/54/NCT02674854/SAP_001.pdf